CLINICAL TRIAL: NCT06176495
Title: Empowering Patients With Diabetes and Their Family Members: Assessing the Impact of Free Informative Mobile Messages
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Najla El Lakkis, Specialist in Family Medicine; Specialist in Occupational Medicine; Clinical Associate in Family Medicine, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SBS-2023-0225
Record Dates: First submitted 2023-11-21; First posted 2023-12-19 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Family Member Caregivers; Education; Educational text messages; WhatsApp
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients with Diabetes and Family Member Caregivers who will receive no text messages over the designated period of the designated
- Intervention Group (Other): Patients with Diabetes and Family Member Caregivers who will receive Educational Text Messages via WhatsApp over the designated period of the intervention
  Interventions: Diagnostic Test: Educational Text Messages

INTERVENTIONS:
Diagnostic Test: Educational Text Messages — The educational content will be targeted about Diabetes Education and will be guideline based with what complies to the standards of care instituted by the American Diabetes Association.
  They text messages will comprise content related to general diabetes knowledge, diabetes management and control, coping with diabetes, and guidance on adopting a healthy lifestyle.
  Arms: Intervention Group

SUMMARY:
This is a Randomized Control Trial aiming at investigating the feasibility and effectiveness of a WhatsApp-based informative intervention on Diabetes Mellitus care in Lebanon and exploring the impact of this intervention on various aspects of Diabetes management and patient outcomes.

Family member caregivers will be also included in this interventional study as the research investigators opt to evaluate their DM related knowledge, personal health practices, their involvement in the care of patients with diabetes, and their impact on the patients' diabetes control before and after the intervention.

DETAILED DESCRIPTION:
Participants with diabetes will be equally and randomly divided into an intervention group (patients with diabetes and their designated family member) of individualized WhatsApp groups which will include each participant individually and the study coordinator to protect their privacy; regular, 4-5 diabetes educational messages a week for a total of 12 weeks will be sent by noon (around 12 pm) to the intervention group participants. The other group, control group, will receive no text messages throughout this period. After 3 months, participants of the intervention group (patients with diabetes and their family members) will be asked to fill in a postintervention knowledge and practices questionnaire to delineate any marked differences in the context of knowledge and health behaviors. All participants with diabetes of both groups will be asked to recheck the previously noted clinical and laboratory parameters at 12 weeks to evaluate for any changes particularly among the intervention group who will also be asked to fill out a postintervention survey. After 6 months, all patients with diabetes will be asked to recheck their clinical and laboratory values again and members of the intervention group will be asked to fill in the practices section questionnaire again.

This research will additionally include Family Members of patients with diabetes who are involved in their care (cooking, aiding in management, securing/delivering medications, etc.). Family Member Caregivers of participants will be designated/noted by the participants who have diabetes themselves, and they will be included in the study based on their willingness to take part of the study. They will also be sorted into either a control or an intervention group in accordance with which group their relative with diabetes was sorted into, for example, if the patient with diabetes will be designated to be a part of the intervention group, this means that the family member caregiver participant will also be allocated to the intervention group. Our aim is to evaluate their DM related knowledge, personal health practices, their involvement in the care of patients with diabetes, and their impact on the patients' diabetes control before and after the intervention.

One point to note as well is that to ensure equality among groups and for the benefit of the control group participants, the research investigators will be sharing with them the content of the text messages originally shared with the participants of the intervention group by the End of the study.

ELIGIBILITY:
Inclusion Criteria for Participants with Diabetes:

* Adult patients 18 years or older
* Patients with an established DM diagnosis
* Patients with a recent HbA1c level with no recent changes in treatment regimen
* Recent HbA1c > 7 but less than 9
* Patients who are on oral antidiabetic medications or basal insulin (intermediate, long acting, ultra long acting insulin)
* Patients who are adherents to the American University of Beirut Health Insurance Plan (AUB-HIP)
* Patients who have visited the Family Medicine Primary Care Clinics at American University of Beirut Clinics in the past 12 months.
* Patients with smart mobile phones and/or access to WhatsApp services
* Patients who can speak and read Arabic or English or live with someone who can read for them
* Patients with available family members involved in their care (e.g. cooking, aiding in management, securing/delivering medications, having the patient medically insured, etc.).
* Willingness to participate in the study

Exclusion Criteria for participants with Diabetes:

* Young patients below 18 years
* Patients who are on non basal insulin/bolus therapy
* Adults with cognitive impairment
* Adults with functional dependence and no assisting family member or caregiver
* Pregnant and Postpartum patients
* Patients with terminal or critical diseases (e.g., cancer; advanced heart, lung, liver, and kidney disease; Human immunodeficiency virus infection and Acquired immune deficiency syndrome and etc.)
* Patients with severe hearing or visual impairment
* Patients who can't read or have difficulty reading and do not live with someone who can read for them
* Patients who will have any of their medications modified throughout the study process will be excluded from the study as well
* Patients with a positive depression (PHQ 2) and/or anxiety (GAD 2) screening results who will be asked to follow up with their primary physician

Inclusion Criteria for Family Member Caregivers:

* Age 18 years or older
* Designated or selected by the participating patient with diabetes.
* Not diagnosed with DM
* Can read and write
* No visual or hearing impairments
* Involved in the participant's diabetes or general care and has an influence on the participant's lifestyle behaviors or medical insurance (e.g. cooking, aiding in management, securing/delivering medications, having the patient medically insured, etc.).
* Access to the WhatsApp service
* Willingness to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Percentage change in glycemic control determined by HbA1C (in percent) in participants with diabetes pre and post intervention. | at 3 and 6 months interval
  To determine the effectiveness of diabetes tailored text messages on glycemic control in patients with diabetes mellitus, Percentage change in glycemic control determined by HbA1C (in percent) in participants with diabetes pre and post intervention will be assessed.

SECONDARY OUTCOMES:
Change in knowledge before and after the intervention (in percentage) | at 3 and 6 months interval
  Assessment of the change in percentage of knowledge in both the patients' and family members' that will be assessed based on the questionnaire that is to be filled before and after the intervention.
  Chi-squared test will be utilised with a p-value of ≤ 0.05 being considered as statistically significant.
Changes in Daily Health Practices pre and post intervention (in percentage) | at 3 and 6 months interval
  the participants daily health practices will be assessed using a designed questionnaire. the changes in health practices will be assessed pre and post intervention using delta percentage.
  Chi-squared test will be utilised with a p-value of ≤ 0.05 being considered as statistically significant.
Percentage change in weight (in Kg), height (in meters) and BMI (Kg/m2) pre and post intervention | At 3 and 6 months interval
  Percentage change in weight (in kg), height ( in meters) and BMI (in Kg/m2) pre and post intervention in participants with diabetes
Percentage change in fasting sugar (mg/dl) pre and post intervention among participants with diabetes | At 3 and 6 months interval
  Percentage change in fasting sugar (mg/dl) pre and post intervention among participants with diabetes
Percentage change in lipid profile composed of Total Cholesterol, LDL, HDL and Triglycerides ( all in mg/dl) among participants with diabetes pre and post intervention | At 3 and 6 months interval
  Percentage change in lipid profile composed of Total Cholesterol, LDL, HDL and Triglycerides ( all in mg/dl) among participants with diabetes pre and post intervention
Percentage change in systolic and diastolic blood pressure (in mmHg) in participants with diabetes pre and post intervention | At 3 and 6 months interval
  Percentage change in systolic and diastolic blood pressure (in mmHg) in participants with diabetes pre and post intervention
Assessment of Changes in Depression Screening score (in percentage pre and post intervention) | At 3 and 6 months interval
  Changes in patients' depression screening score pre and post intervention using the PHQ 2 scaled score. This will be reflected in percentage (pre and post intervention) to reflect the changes in the participants' mood. Chi-squared test will be utilised with a p-value of ≤ 0.05 being considered as statistically significant.
  For the PHQ-2, the score ranges from 0-6. A score of 3 is considered as the optimal cut point when using the PHQ-2 to screen for depression. If the score is 3 or greater, major depressive disorder is likely.
Assessment of Changes in Anxiety Screening score (in percentage pre and post intervention) | At 3 and 6 months interval
  Changes in patients' anxiety screening score pre and post intervention using the GAD 2 scaled score. This will be reflected in percentage (pre and post intervention) to reflect the changes in the participants' mood. Chi-squared test will be utilised with a p-value of ≤ 0.05 being considered as statistically significant.
  For the GAD-2, the score ranges from 0-6. A score of 3 is considered as the optimal cut point when using the GAD-2 to screen for generalised anxiety. If the score is 3 or greater, generalised anxiety is likely.

CONTACTS AND LOCATIONS:
Overall Officials: Najla El Lakkis, FAM MED, Principal Investigator — American University of Beirut Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Mutawaa KA, Farghaly AH, Nasir R, Loares AM, Skaroni I, Al-Thani M, Abou-Samra AB. Level of knowledge, attitude and practice towards diabetes among nationals and long-term residents of Qatar: a cross-sectional study. BMJ Open. 2022 Feb 16;12(2):e052607. doi: 10.1136/bmjopen-2021-052607. PMID 35172997
- [Result] Abaza H, Marschollek M. SMS education for the promotion of diabetes self-management in low & middle income countries: a pilot randomized controlled trial in Egypt. BMC Public Health. 2017 Dec 19;17(1):962. doi: 10.1186/s12889-017-4973-5. PMID 29258499
- [Result] Ernawati U, Wihastuti TA, Utami YW. Effectiveness of diabetes self-management education (DSME) in type 2 diabetes mellitus (T2DM) patients: Systematic literature review. J Public Health Res. 2021 Apr 14;10(2):2240. doi: 10.4081/jphr.2021.2240. PMID 33855427
- [Result] Karaoui LR, Deeb ME, Nasser L, Hallit S. Knowledge and practice of patients with diabetes mellitus in Lebanon: a cross-sectional study. BMC Public Health. 2018 Apr 20;18(1):525. doi: 10.1186/s12889-018-5416-7. PMID 29678148
- [Result] Sahin C, Courtney KL, Naylor PJ, E Rhodes R. Tailored mobile text messaging interventions targeting type 2 diabetes self-management: A systematic review and a meta-analysis. Digit Health. 2019 Apr 22;5:2055207619845279. doi: 10.1177/2055207619845279. eCollection 2019 Jan-Dec. PMID 31041110
- [Result] Bin Abbas B, Al Fares A, Jabbari M, El Dali A, Al Orifi F. Effect of mobile phone short text messages on glycemic control in type 2 diabetes. Int J Endocrinol Metab. 2015 Jan 1;13(1):e18791. doi: 10.5812/ijem.18791. eCollection 2015 Jan. PMID 25745493
- [Result] Omar MA, Hasan S, Palaian S, Mahameed S. The impact of a self-management educational program coordinated through WhatsApp on diabetes control. Pharm Pract (Granada). 2020 Apr-Jun;18(2):1841. doi: 10.18549/PharmPract.2020.2.1841. Epub 2020 May 3. PMID 32477434
- See also: statistical figures — https://idf.org/about-diabetes/facts-figures/
- See also: statistical figures — https://pubmed.ncbi.nlm.nih.gov/32141596/
- See also: statistical figures — https://apps.who.int/gho/data/view.main.NCDRGLUCAv?lang=en%5D
- See also: SMS education for the promotion of diabetes self-management in low & middle income countries: a pilot randomized controlled trial in Egypt — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5735794/
- See also: Effectiveness of diabetes self-management education (DSME) in type 2 diabetes mellitus (T2DM) patients: Systematic literature review — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8129774/
- See also: Educating diabetic patients through an SMS intervention: a randomized controlled trial at a Brazilian public hospital — https://www.scielo.br/j/aem/a/VCBKnRL6km3qjGsf3LbFDFg/?lang=en
- See also: Knowledge and practice of patients with diabetes mellitus in Lebanon: a cross-sectional study — https://pubmed.ncbi.nlm.nih.gov/29678148/
- See also: Level of knowledge, attitude and practice towards diabetes among nationals and long-term residents of Qatar: a cross-sectional study (With KAP Questionnaire) — https://pubmed.ncbi.nlm.nih.gov/35172997/
- See also: Disease-related distress, self-care and clinical outcomes among low-income patients with diabetes — https://jech.bmj.com/content/68/6/557.long
- See also: Family-Centered Diabetes Care for Better Glycemic Outcomes of Outpatients in Rural Areas — https://www.intechopen.com/chapters/75367
- See also: Tailored mobile text messaging interventions targeting type 2 diabetes self-management: A systematic review and a meta-analysis — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6481002/
- See also: Effect of Mobile Phone Short Text Messages on Glycemic Control in Type 2 Diabetes — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4338653/
- See also: The impact of a self-management educational program coordinated through WhatsApp on diabetes control — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7243744/